CLINICAL TRIAL: NCT00710671
Title: Psychosocial Needs of HIV+ Young Men Who Have Sex With Men (YMSM)
Brief Title: Psychosocial Needs of YMSM
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: ATN 070
Record Dates: First submitted 2008-07-02; First posted 2008-07-04 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-02

CONDITIONS: HIV+ YMSM
Keywords: HIV positive; YMSM; risk factors; coping; identity development; psychosocial needs
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Phase 1: Male, HIV+ participants from ages 16-24 who have had sex with another male in the past year and acquired HIV behaviorally. Participants will be drawn from four participating AMTU sites.
- Phase 2: Male, HIV+ participants from ages 16-24 who have had sex with another male in the past year and acquired HIV behaviorally. Participants will be drawn from all fifteen AMTU sites.

SUMMARY:
The proposed study will use both qualitative and quantitative research methods (mixed methods) to gather data that will support the eventual development of interventions for young men who have sex with men (YMSM) living with behaviorally acquired HIV infection. The overall goal of the study is to gain an understanding of the psychosocial/developmental needs of YMSM by focusing on two critical developmental issues-identity development and future life goals.

ELIGIBILITY:
Inclusion Criteria:

Potential participants must meet all of the following inclusion criteria in order to participate in the study:

* Biologically male at birth and identifies as male at time of study participation;
* HIV-infected as documented by medical record review or verbal verification with referring professional;
* Between the age of 16 years, 0 days to 24 years, 364 days at the time of informed consent/assent;
* HIV infection occurred through sexual or substance use behavior of the participant;
* Ability to understand both written and spoken English; and
* History of at least one sexual encounter involving either anal or oral penetration (either receptive or insertive) with a male partner during the 12 months prior to enrollment.

Exclusion Criteria:

* Acquired HIV through perinatal infection;
* Transfusion acquired HIV infection;
* Presence of serious psychiatric symptoms (active hallucinations, thought disorder) that would impair participants' ability to complete the study measures;
* Visibly distraught (suicidal, homicidal, exhibiting violent behavior); or
* Intoxicated

Ages: 16 Years to 24 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Male, HIV+ participants from ages 16-24 who have had sex with another male in the past year and accquired HIV behaviorally.
Sampling Method: Non-Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2008-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
An understanding of the most salient risk factors/stressors and resistance factors/coping mechanisms that impact healthy identity development among YMSM living with HIV. | To be determined in analysis
An understanding of the association between ethnic identity, sexual identity, and identity as a young man living with HIV and the health behaviors of substance use, sexual activity, and adherence to healthcare among YMSM living with HIV. | To be determined in analysis
An understanding of the most salient risk factors/stressors and resistance factors/coping mechanisms that negatively impact the future life goals of YMSM living with HIV. | To be determined in analysis
Identification of additional psychosocial/developmental needs of YMSM living with HIV (in addition to healthy identity development and future life goals). | To be determined in analysis
Development of recommendations for interventions aimed at facilitating healthy identity development, constructing future life goals, and addressing additional psychosocial/developmental needs among YMSM living with HIV. | To be determined in analysis

CONTACTS AND LOCATIONS:
Overall Officials: Gary W Harper, Study Chair — Adolescent Trials Network
Locations (14):
- United States (14):
  - Children's Hopsital of Los Angeles, Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Diagnostic and Teatment Center, Fort Lauderdale, Florida
  - University of Miami, Miami, Florida
  - University of South Florida College of Medicine, Tampa, Florida
  - John Stroger Jr. Hospital of Cook County, Chicago, Illinois
  - Children's Memorial Hospital, Chicago, Illinois
  - Tulane Medical Center, New Orleans, Louisiana
  - University of MD School of Medicine, Baltimore, Maryland
  - Mount Sinai Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee